CLINICAL TRIAL: NCT01497236
Title: Effectiveness of Nutritional Supplementation (RUTF and Multi Micronutrient) in Preventing Malnutrition in Children 6-59 Months With Infection (Malaria, Pneumonia, Diarrhoea), a Randomized Controlled Trial in Kaabong, Karamoja, Uganda
Brief Title: Effectiveness of Nutritional Supplementation in Preventing Malnutrition in Children With Infection in Karamoja, Uganda
Acronym: MSF-nutcon03
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medecins Sans Frontieres, Spain (Other)
Responsible Party: Principal Investigator, Nuria Salse, Nutrition Advisor MSF Spain, Medecins Sans Frontieres, Spain
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MSF-nutcon03
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Child Malnutrition; Infant Morbidity
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Experimental: Ready to Use Terapeutic Food (RUTF) (Experimental)
  Interventions: Dietary Supplement: Dietary Supplement: Nutrition supplement with RUTF or MNP
- Multi Micronutrient Powder (MNP) (Experimental)
  Interventions: Dietary Supplement: Dietary Supplement: Nutrition supplement with RUTF or MNP
- no supplement (No Intervention)

INTERVENTIONS:
Dietary Supplement: Dietary Supplement: Nutrition supplement with RUTF or MNP — 14 days nutritional supplementation with either
  * a fortified high quality food(RUTF), 1 sachet/day, 500 kcal and multi micronutrients
  * a multi micronutrient powder (MNP), 2 sachets per day, no calories, twice recommended daily intake
  * a placebo (to MNP), 2 sachets per day , no calories, no micronutrients, containing micronutrient carrier
  Other Names: Other Names:; RUTF: Nutriset; MNP: MixMe, DSM; Placebo: DSM
  Arms: Experimental: Ready to Use Terapeutic Food (RUTF); Multi Micronutrient Powder (MNP)

SUMMARY:
The purpose of this study is to determine whether 14 days nutritional supplementation with Ready to use therapeutic Food (RUTF) or micronutrients alone to children having an infection will prevent malnutrition and reduce the frequency of morbidity.

DETAILED DESCRIPTION:
similar to MSF-nutcon 03 : NCT01154803

ELIGIBILITY:
Inclusion Criteria:

* 6 to 59 months of age
* Not malnourished
* Diagnosis of malaria and/or diarrhoea and/or LRTI
* Intending to remain in area for the duration of the 6 month follow-up
* Living within approximately 60 minutes walking distance from the clinic
* Informed consent from a guardian*

Exclusion Criteria:

* Child is exclusively breastfeeding
* Child is severely malnourished
* Presence of 'General Danger Signs'
* Presence of severe disease (including severe malaria, severe LRTI, severe diarrhoea)
* Needing hospitalisation for any reason
* Known history of allergy to the nutritional supplementation
* Having a sibling enrolled in the study*

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2202 (Actual)
Dates: Start 2011-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
"negative nutritional outcome" of a child | 6 months follow-up
  The incidence of a negative nutritional outcome will be defined in two different ways according to the baseline nutritional status.
  i) for children with no malnourishment at time of entry into study, "negative nutritional outcome" is defined as progression to moderate or severe malnourishment ii) for children with moderate malnourishment at time of entry into study, "negative nutritional outcome" is defined as loss of ³10% of baseline weight or progression to severe malnourishment, whichever is reached first

SECONDARY OUTCOMES:
Number of new events of a study disease | 6 months
  study disease: malaria, diarrhoea, and LRTI

CONTACTS AND LOCATIONS:
Overall Officials: Nuria Salse, Principal Investigator — MSF Spain
Locations (1):
- Kaabong Hospital, Kaabong, Karamoja District, Uganda

REFERENCES:
- [Derived] van der Kam S, Roll S, Swarthout T, Edyegu-Otelu G, Matsumoto A, Kasujja FX, Casademont C, Shanks L, Salse-Ubach N. Effect of Short-Term Supplementation with Ready-to-Use Therapeutic Food or Micronutrients for Children after Illness for Prevention of Malnutrition: A Randomised Controlled Trial in Uganda. PLoS Med. 2016 Feb 9;13(2):e1001951. doi: 10.1371/journal.pmed.1001951. eCollection 2016 Feb. PMID 26859481